CLINICAL TRIAL: NCT05708430
Title: Tolerance of Intra-articular Injection Autologous Stromal Vascular Fraction for the Treatment of Rhizarthrosis
Acronym: FVS-RHIZA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/0419/HP
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Rhizarthrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SVF injection (Experimental): Intra-articular injection of autologous cells from the stromal vascular fraction derived from adipose tissue
  Interventions: Drug: SVF injection into wrist

INTERVENTIONS:
Drug: SVF injection into wrist — Intra-articular injection of autologous cells from the stromal vascular fraction derived from adipose tissue

SUMMARY:
Rhizarthosis is a common disease in the population (15%). It has a major impact on the function of the hand since it compromises the pollicidigitales claws and all gripping functions with the thumb. However, no curative medical treatment exists to date. The treatment is initially based on a symptomatic approach: analgesics, non-steroidal anti-inflammatories, immobilization orthoses or even intra-articular injections of corticosteroids or hyaluronic acid. When it is exceeded, surgical treatment is considered. This is also not a curative treatment. Indeed, the 3 types of main interventions proposed (arthrodesis, arthroplasty or trapezectomy) each have significant consequences for the patient: stiffness for the arthrodesis, risk of dislocation or failure of the material for the prosthesis, long consequences for the trapezectomy. , or potential complications of surgery.

Stem cell-based therapies, in particular cells of the stromal vascular fraction derived from adipose tissue (FVS), are promising in various indications, including osteoarthritis of the knee. Autologous FVS is readily accessible by standard liposuction, with FVS isolated from adipose tissue by centrifugation. A safe and well-tolerated source of cells with angiogenic, anti-inflammatory, immunomodulatory and regenerative properties, its safety has been demonstrated in particular during phase 1 trials. Our objective is to assess the tolerance of an injection of FVS into the trapezio-metacarpal joint, when standard medical treatment has failed, and the rhizarthrosis has become painful enough to be eligible for surgery. Due to its immunomodulatory and cartilage regeneration properties, this injection would be performed to offer a less invasive and possibly curative treatment instead of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Rhizarthrosis DELL stage 1 to 3 (see appendix 1)
* Symptomatic medical treatment for a period of at least 6 months (analgesic, orthosis, anti-inflammatory, etc. or intra-articular infiltration of the trapezio-metacarpal joint) which has become ineffective (surgical stage)
* EVA pain ≥ 4
* Quick Dash or PRWHE ≥ 20/100 (see Appendices 2 and 3)
* Affiliation to a social security scheme
* Person who has read and understood the information letter and signed the consent form

Exclusion Criteria:

* History of intra-articular injection of the trapezio-metacarpal (corticoid or hyaluronic acid) in the last 6 months
* Body Mass Index < 18 kg/m2
* Contraindication to general or local anesthetics including XYLOCAINE 10 mg/mL ADRENALINE 0.005 mg/mL, solution for injection
* Contraindication to sedation or general anesthesia (left to the discretion of the anesthesiologist)
* Contraindication to liposuction (eg bleeding disorder)
* Documented severe allergy to conventional antibiotics such as β-lactams, cyclins, macrolides, quinolones, aminoglycosides, etc…
* Known hypersensitivity to human albumin or to any of the excipients (VIALEBEX 200 g/L, solution for infusion)
* A general or local infection near the sampling or injection sites
* Any surgery scheduled over the duration of the study of the hand (carpal tunnel type operation) or upper limb that may have an impact on the assessment of pain and/or functional indices
* Persons on immunosuppressants: corticosteroid therapy > 10 mg/d, methotrexate > 25 mg/week, mycofenolate mofetil > 3 grams/d, azathioprine > 200 mg/d and intravenous cyclophosphamide and any biotherapy in the 90 days preceding the medical visit. inclusion
* Congenital or acquired immune deficiency
* Prescription of a new systemic treatment that may influence the condition of the hand (vasodilator or immunosuppressant) in the 90 days preceding inclusion
* Persons infected with HIV, HCV, HBV, HTLV and syphilis
* Contraindication to MRI, (eg, due to presence of pacemakers or other incompatible foreign material or claustrophobia)
* Contraindication to the injection of gadolinated contrast product (gadolinium) for performing MRI (history of hypersensitivity to gadolinated contrast products)
* Active COVID-19 infection (PCR positive)
* Any cardiovascular, metabolic, endocrine, psychiatric or cancerous pathology in uncontrolled evolution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the number of treatment-attributable Grade ≥ 3 adverse reactions occurring over a 6-month period after intra-articular injection of FVS. | 6 months
  The primary endpoint is the number of treatment-attributable Grade ≥ 3 adverse reactions occurring over a 6-month period after intra-articular injection of FVS.

IPD SHARING:
Plan to Share IPD: No